CLINICAL TRIAL: NCT00078845
Title: Phase II Trial Of Subcutaneous Amifostine For Reversal Of Persistent Paclitaxel-Induced Peripheral Neuropathy
Brief Title: Amifostine in Treating Peripheral Neuropathy Caused by Paclitaxel in Patients With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000330006; MDA-CCC-0223; MDA-CCC-0203; MDA-2003-0789
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer; Lung Cancer; Neurotoxicity; Ovarian Cancer; Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neurotoxicity; unspecified adult solid tumor, protocol specific; recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; limited stage small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent ovarian epithelial cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Neurotoxicity Syndromes; Ovarian Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Ovarian Epithelial | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amifostine (Experimental): 500 mg subcutaneous three times a week on Monday, Wednesday and Friday for 4 weeks.
  Interventions: Drug: Amifostine

INTERVENTIONS:
Drug: Amifostine — 500 mg three times a week.
  Other Names: amifostine trihydrate

SUMMARY:
RATIONALE: Amifostine may be effective in reducing pain, numbness, tingling, and other symptoms of peripheral neuropathy.

PURPOSE: This phase II trial is studying how well amifostine works in reducing pain, numbness, tingling, and other symptoms of peripheral neuropathy in patients who have received paclitaxel for solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the percentage of patients with solid tumors who have persistent paclitaxel-induced peripheral neuropathy who benefit, defined as a decrease of at least 20% on their FUNCTIONAL ASSESSMENT OF CANCER THERAPY/ GYNECOLOGIC ONCOLOGY GROUP NEUROTOXICITY (FACT/GOG-Ntx) FACT-GOG-NTX score, from treatment with subcutaneous amifostine.
* Determine whether there is sufficient evidence of reversal activity of this drug in these patients to justify a phase III study.

Secondary

* Compare the acute toxic effects of this drug administered subcutaneously in these patients vs IV administrations of this drug historically and/or during the GOG-0192 study.
* Determine the capability of the Weinstein Enhanced Sensory Test to provide objective, quantitative evidence for improvement in patients who have subjective improvement as self-reported on the FACT-GOG-NTX scale.
* Determine whether any benefit in patients treated with this drug is transient or lasts at least 8 weeks.

OUTLINE: This is an open-label, multicenter study.

Patients receive amifostine subcutaneously three times weekly for 4 weeks in the absence of symptom progression or unacceptable toxicity. Patients achieving a complete or partial response receive an additional 4 weeks of therapy.

Neuropathy symptoms are assessed using the FACT-GOG-NTX questionnaire administered at baseline, weekly during therapy, and at 12 weeks and the Weinstein Enhanced Sensory Test administered at baseline and at 4, 8, and 12 weeks.

Patients are followed at 12 weeks.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 10-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a solid tumor, including, but not limited to the following:

  * Ovarian cancer
  * Lung cancer
  * Prostate cancer
  * Breast cancer
* Previously treated with paclitaxel
* Peripheral neuropathy (e.g., numbness, tingling, and/or pain in distal extremities) believed to be caused by paclitaxel only or the combination of paclitaxel and carboplatin

  * At least 18 out of 44 on the FACT-GOG-NTX scale
  * Persistent neuropathy for at least 2, but no more than 12 months after chemotherapy
  * Not improving
* No other possible cause of neuropathy (e.g., alcoholism, diabetes, or peripheral vascular disease)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Karnofsky 50-100%

Life expectancy

* More than 2 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL
* Calcium ≥ lower limit of normal

Cardiovascular

* See Disease Characteristics
* No prior cerebrovascular accident

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other significant comorbid medical condition that would preclude study participation
* No known sensitivity to aminothiol compounds

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior cisplatin
* No chemotherapy during and for at least 3 months after study participation

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent monoamine oxidase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Neurotoxicity secondary to cancer therapy as measured by FACT-GOG-NTX scale | 12 weeks
  11-item FACT/GOG-NTX questionnaire completed weekly following chemotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Forman, MD, Study Chair — M.D. Anderson Cancer Center
Locations (15):
- United States (15):
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - Christus St. Frances Cabrini Center for Cancer Care, Alexandria, Louisiana
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin